CLINICAL TRIAL: NCT02800031
Title: The Diagnostic Value Of International Ovarian Tumour Analysis (IOTA) Simple Rules Versus the Pattern Recognition Method In Differentiating Between Malignant And Benign Adnexal Masses
Brief Title: IOTA Versus Pattern Recognition Method in Diagnosis of Ovarian Masses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Dina Mohamed Refaat Dakhly, Assistant Professor Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: HJ200516
Record Dates: First submitted 2016-04-26; First posted 2016-06-15 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Gynecology

STUDY DESIGN:
Masking Description: Level-II Transvaginal ultrasonography will be done by the principle investigator (who is unaware about the recognition pattern method) to confirm the presence of the ovarian mass and measure its size and to apply the IOTA simple rules on it (complimentary transabdominal ultrasound might be done for huge pelvi-abdominal masses originating from the ovary).
  Level-III ultrasound will be done by expert ultrasound operator (who is blinded to the results of IOTA simple rules assessment of the examined mass) to classify the mass (either benign or malignant) using the pattern recognition method.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Participants (Experimental): * Level-II Transvaginal ultrasonography will be done by the principle investigator (who is unaware about the recognition pattern method) to confirm the presence of the ovarian mass and measure its size and to apply the IOTA simple rules on it (complimentary transabdominal ultrasound might be done for huge pelvi-abdominal masses originating from the ovary).
  * Level-III ultrasound will be done by expert ultrasound operator (who is blinded to the results of IOTA simple rules assessment of the examined mass) to classify the mass (either benign or malignant) using the pattern recognition method.
  * Plan of management for each patient will be based solely on the findings of pattern recognition and the patient's wishes.
  * Exploratory laparotomy for excision of the ovarian mass either by ovarian Cystectomy or oophorectomy.
  * All specimens will be examined histopathologically.
  Interventions: Device: Transvaginal ultrasonography

INTERVENTIONS:
Device: Transvaginal ultrasonography

SUMMARY:
To compare between the efficacy of IOTA simple rules and pattern recognition method in the differentiating between benign and malignant adnexal masses

ELIGIBILITY:
Inclusion Criteria:

* Ovarian mass more than 5 cm in size (confirmed by transvaginal or transabdominal ultrasonography in gynecology clinic)
* The patient is candidate for abdominal exploration for ovarian Cystectomy or oophorectomy.

Exclusion Criteria:

* Complicated ovarian masses.
* Unfit for surgery.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2016-04; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
comparing the sensitivity of the IOTA versus the Pattern recognition in diagnosing the different types of ovarian masses | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Dina MR Dakhly, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr el aini hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dakhly DMR, Gaafar HM, Sediek MM, Ibrahim MF, Momtaz M. Diagnostic value of the International Ovarian Tumor Analysis (IOTA) simple rules versus pattern recognition to differentiate between malignant and benign ovarian masses. Int J Gynaecol Obstet. 2019 Dec;147(3):344-349. doi: 10.1002/ijgo.12970. Epub 2019 Sep 26. PMID 31520402